CLINICAL TRIAL: NCT01256944
Title: To Study Polycystic Ovary Syndrome in Taiwanese Women
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, MD, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-99041
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Syndrome; Cardiovascular Disease
Keywords: PCOS; DM; Hypertension; CVD
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: The normal reproductive-aged women
- PCOS: Women who met the 2003 Rotterdam criteria, which require a minimum of two of the following three criteria:
  1. Oligo- or anovulation
  2. Clinical and/or biochemical signs of hyperandrogenism
  3. Polycystic ovaries and exclusion of other etiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome)

SUMMARY:
Polycystic ovary syndrome (PCOS) is an extremely common disorder in women of reproductive age. Diagnosis of PCOS is principally based on clinical and physical findings. Diagnostic criteria and PCOS definitions used by clinicians and researchers are almost as heterogeneous as the syndrome. Of those diagnosed with PCOS using the 2003 Rotterdam criteria, 61% fulfilled 1990 NIH criteria for unexplained hyperandrogenic chronic anovulation. The patient populations with the new phenotypes had less severe ovulatory dysfunction and less androgen excess than patients diagnosed using the 1990 NIH criteria. These findings might be common across all female populations with PCOS, whether in Oriental or Occidental countries. Data for clinical hyperandrogenism indicated that the prevalence of hirsutism in Taiwanese PCOS women is lower than that for Caucasians/Western women.

The extent of metabolic abnormalities in women with PCOS may vary with phenotype, age and ethnicity. Obesity represents a major risk factor for metabolic syndrome and insulin resistance. Approximately 40-50% of all women with PCOS are overweight or obese. Obese subjects with PCOS had a higher risk of developing oligomenorrhea, amenorrhea and biochemical hyperandrogenemia than non-obese women with PCOS. Moreover, obese women with PCOS had significantly more severe insulin resistance, lower serum LH levels, and lower LH-to-FSH ratios than non-obese women with PCOS. PCOS women in Taiwan presented with higher LH-to-FSH ratio and lower insulin resistance than PCOS women in Western Countries. However, the average body mass index (BMI) was significantly lower in Taiwanese PCOS women than Western women, which might partially explain the difference between these two populations in terms of clinical and biochemical presentations.

To further document the ethnic variation between women with PCOS in Taiwan and Western, the effect of obesity on the diagnosis and clinical presentations of PCOS-related syndromes should not be neglected in future studies. Therefore, the investigators plan to do this prospective study for evaluation the clinical and biochemical presentation of Taiwanese women with PCOS.

DETAILED DESCRIPTION:
1. Method

1. This study was approved by the Institutional Review Board of the Wan Fang Medical Center at Taipei Medical University (WF99041, approved August 2010) and performed at the Reproductive Endocrinology Clinic at the Wan Fang Medical Center from 31 August 2010 to 31 August 2011. The following women were excluded: (i) women who had been diagnosed with hyperprolactinemia, hypogonadotropic hypogonadism, premature ovarian failure, congenital adrenal hyperplasia, androgen-secreting tumor,Cushing's syndrome, disorders of the uterus and chromosomal anomalies; (ii) women who were less than three years past menarche or who were older than 45 years; (iii) women who received hormones or medication for major medical diseases (diabetes or cardiovascular disease); and (iv) women who had had ovarian cysts or ovarian tumors identified by ultrasonographic examination.
2. Statistical analysis: We used chi-squared and Fisher's exact tests to perform categorical comparisons and ANOVA to compare the continuous variables. The means of more than two groups were compared using one-way ANOVA and post hoc Dunnett's t-test with equal variances not assumed.

ELIGIBILITY:
Inclusion Criteria:

* women at reproductive age
* women with PCOS and women without PCOS.

Exclusion Criteria:

* young women who had their menarche less than 3 years
* women older than 45 years old, Amenorrhea of menopause, hyperglycemia, hyperthyroidism, hypothyroidism, heart failure, lung failure, renal failure, anemia, dystrophy, gonitis.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: The normal women
Period: Overall Study
Arm/Group | Control | PCOS
Started | 70 | 220
Completed | 70 | 220
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PCOS | Total
Number analyzed (Participants) | 70 | 220 | 290
Age, Continuous [Mean (Standard Deviation); unit: years old] | 28.3 (4.4) | 26.9 (5.8) | 27.68 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 220 | 290
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 70 | 220 | 290

OUTCOME MEASURES:

1. Primary Outcome: Total Testosterone
Description: Using serum total testosterone to represent the severity of hyperandrogenism.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
nmol/L | 1.5 (0.6) | 2.9 (1.2)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: BMI
Description: BMI categorization was based on the WHO Asia-Pacific classification for obesity, which was defined as BMI ≧ 25 kg/m2(WHO: Obesity: preventing and managing the global epidemic. Geneva: WHO; 2000).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
kg/m2 | 23.4 (5.2) | 25.9 (6.1)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

3. Primary Outcome: Fasting Insulin
Description: A fasting serum insulin level of greater than the upper limit of normal for the assay used (approximately 60 pmol/L) is considered evidence of insulin resistance.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: μIU/ml
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
μIU/ml | 8.3 (5.7) | 13.5 (14.5)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

4. Primary Outcome: Fasting Glucose
Description: Fasting blood sugar (FBS) measures blood glucose after you have not eaten for at least 8 hours. It is often the first test done to check for prediabetes and diabetes.
  World Health Organization 2006 diagnostic criteria for diabetes were employed (fasting plasma glucose ≥7.0 mmol/L or two hour plasma glucose ≥11.1 mmol/L).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 5.0 (1.0) | 5.1 (0.8)

5. Primary Outcome: Two Hour Glucose
Description: 2-hour postprandial blood sugar measures blood glucose exactly 2 hours after you start eating a meal. This is not a test used to diagnose diabetes.
  World Health Organization 2006 diagnostic criteria for diabetes were employed (fasting plasma glucose ≥7.0 mmol/L or two hour plasma glucose ≥11.1 mmol/L).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 5.4 (1.1) | 6.4 (2.5)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

6. Primary Outcome: Homeostasis Model Assessment Insulin Resistance Index (HOMA-IR)
Description: HOMA-IR = [fasting insulin (in μIU/mL) × fasting glucose (in mg/dL)]/405.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
unitless | 1.9 (1.3) | 3.2 (3.7)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

7. Primary Outcome: Cholesterol
Description: Hypercholesterolemia was defined as >6 mmol / L.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 4.5 (0.8) | 4.9 (0.9)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

8. Primary Outcome: Triglycerides
Description: Abnormal serum triglycerides defined as ≥ 1.7 mmol/L
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 0.8 (0.5) | 1.1 (0.9)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

9. Primary Outcome: HDL
Description: Metabolic syndrome was defined (2005 National Cholesterol Education Program, Adult Treatment Panel III) as the presence of at least three of the following criteria:
  abdominal obesity (waist circumference >80 cm in women); serumtriglycerides≥1.7 mmol/L; serumHDL<1.3 mmol/L; systolic blood pressure ≥130 mmHg and/or diastolic blood pressure ≥85 mmHg; and fasting plasma glucose ≥7.0 mmol/L.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 1.4 (0.5) | 1.3 (0.4)

10. Primary Outcome: LDL
Description: Lipid profiles, including total cholesterol, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and sex hormone binding globulin (SHBG).
  Abnormal LDL was ≧4.14mmol/L.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | PCOS
Number analyzed (Participants) | 70 | 220
mmol/L | 2.6 (0.6) | 3.0 (0.8)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p < 0.05, ANOVA

11. Primary Outcome: Impaired Glucose Tolerance
Description: Impaired glucose tolerance was defined as two hour glucose levels of 7.8-11.1 mmol/L in the 75 g oral glucose tolerance test. In women with impaired glucose tolerance, the fasting plasma glucose level should be <7 mmol/L.
Time Frame: 1 years
Measure: Number; unit: percentage of participants
Groups:
- Obese With PCOS: BMI categorization was based on the WHO Asia-Pacific classification for obesity, which was defined as BMI ≧ 25 kg/m2(WHO: Obesity: preventing and managing the global epidemic. Geneva: WHO; 2000).
  Women who met the 2003 Rotterdam criteria, which require a minimum of two of the following three criteria:
  1. Oligo- or anovulation
  2. Clinical and/or biochemical signs of hyperandrogenism
  3. Polycystic ovaries and exclusion of other etiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome)
- Obese With Control: BMI categorization was based on the WHO Asia-Pacific classification for obesity, which was defined as BMI ≧ 25 kg/m2(WHO: Obesity: preventing and managing the global epidemic. Geneva: WHO; 2000).
- Non-obese With PCOS: BMI categorization was based on the WHO Asia-Pacific classification for obesity, which was defined as BMI < 25 kg/m2(WHO: Obesity: preventing and managing the global epidemic. Geneva: WHO; 2000).
  Women who met the 2003 Rotterdam criteria, which require a minimum of two of the following three criteria:
  1. Oligo- or anovulation
  2. Clinical and/or biochemical signs of hyperandrogenism
  3. Polycystic ovaries and exclusion of other etiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome)
- Nonb-obese With Control: BMI categorization was based on the WHO Asia-Pacific classification for obesity, which was defined as BMI < 25 kg/m2(WHO: Obesity: preventing and managing the global epidemic. Geneva: WHO; 2000).
Arm/Group | Obese With PCOS | Obese With Control | Non-obese With PCOS | Nonb-obese With Control
Number analyzed (Participants) | 110 | 20 | 110 | 50
percentage of participants | 43 | 25 | 10 | 0
Statistical Analysis 1: Comparison: Non-obese With PCOS vs Nonb-obese With Control; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year 1 month
Arm/Group | Control | PCOS
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/220
Other Adverse Events (participants affected / at risk) | 0/70 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No